CLINICAL TRIAL: NCT00920127
Title: An Investigation of the Safety and Efficacy of Oral AKL1 in Patients Diagnosed With Obstructive Lung Disease
Brief Title: Treatment With AKL1 in Obstructive Airways Disease (The TAKL Study)
Acronym: TAKL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of East Anglia (Other)
Responsible Party: Dr Andrew M Wilson, University of East Anglia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32227/0001/001; EudraCT: 2222 - 222222-22
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Obstructive Lung Disease; Chronic Obstructive Pulmonary Disease; Asthma
Keywords: AKL1; COPD
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: AKL1
- AKL1 (Active Comparator)
  Interventions: Dietary Supplement: AKL1

INTERVENTIONS:
Dietary Supplement: AKL1 — Each dose of AKL1 or placebo will consist of two capsules which will be swallowed twice daily for 8 weeks.
  The morning dose of study medication should be taken at approximately the same time each morning between 7:00 am and 10:00 am and should consist of two 500 mg capsules and then repeated between 7.00 pm and 10 pm.

SUMMARY:
Obstructive airways disease is a very common condition. This condition includes patients with asthma, chronic obstructive pulmonary disease (COPD), emphysema or chronic bronchitis. Some patients with obstructive airways disease have problems with long term breathlessness, wheeze and cough with or without sputum production. Currently the researchers give treatments - usually inhalers - which are designed to open the airways and reduce the breathlessness and wheeze. Despite these available treatments many patients still have continuing symptoms.

Anecdotal clinical evidence suggested that a herbal remedy (called AKL1) has beneficial effects in respiratory conditions, with patients diagnosed as having both asthma and COPD reporting reduced symptoms including breathlessness and cough and reduced frequency of attacks.The purpose of this study is to confirm whether AKL1 does indeed have a meaningful benefit to patients with obstructive airways disease. The researchers will mainly be measuring any effect of AKL by assessing any change in trial subjects' coughs, using a questionnaire, but the researchers will also looking at breathing tests, walking tests, blood and sputum tests.

DETAILED DESCRIPTION:
The outcomes of care for obstructive airways disease in the UK and other countries fail to meet guideline targets, with high levels of avoidable morbidity and avoidable mortality. Obstructive lung disease is an encompassing term for a condition that includes patients with a reversible (asthma) or non reversible (chronic obstructive pulmonary disease) component to their lung function.

AKL1 is a novel pharmaceutical agent derived from a combination of botanical products developed as a treatment for obstructive lung disease (asthma and COPD). The botanical product contains a synthetically-derived phytochemical component of Picrorrhiza kurroa, apocynin, together with standardized extracts of Picrorrhiza kurroa, Zingiber officinale and Ginkgo biloba that have previously been marketed as a health food supplements. Recent evidence suggests that Ginkgo biloba reduces inflammatory (protein kinase C positive ie eosinophils and neutrophils) cells in induced sputum which given in addition to inhaled corticosteroids to asthmatic patients. Anecdotal clinical evidence suggests that the botanical product has significant activity in respiratory conditions, with patients diagnosed as having obstructive lung disease (asthma and COPD) reporting reduced symptoms including breathlessness and cough, reduced frequency of attacks, reduced dependence on bronchodilators and ability to reduce inhaled corticosteroids dose.

We have completed a pilot study investigating the efficacy and safety of AKL1 as 'add-on' therapy for adult patients diagnosed as having obstructive lung disease whose symptoms remained uncontrolled on standard medication. Whilst there was no significant differences in lung function, there were trends to clinical improvements in the patient-centered outcomes e.g. cough, health status and exacerbation frequency. Hence a larger adequately powered study is needed to investigate these outcomes further.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged between 18 to 80 years, inclusive
* The patient has received verbal and written study information, all questions have been answered satisfactorily and a consent form has been personally signed and dated by the patient and the investigator
* A diagnosis of obstructive lung disease (with reference to the - International Primary Care Respiratory Group (IPCRG) Guidelines)(4). This being evidenced as a post bronchodilator ratio of FEV1/FVC < 0.7 at Visit 1 or 2 The patient has a post bronchodilator FEV1 of greater than 40% and less than 80% at Visit 1 or 2
* Patients have a history of regular sputum production (> 3 days per week)
* LCQ score of <17 (higher score indicates improvement).
* A MRC dyspnoea score of 3 or more
* Females must be post menopausal (> 1 year), surgically sterilised or using adequate hormonal contraception, intrauterine device), not breast feeding and have a negative serum pregnancy test
* The patient must have a satisfactory health with the exception of obstructive lung disease as determined by the investigator on the basis of medical history and physical examination
* In the Investigator's judgement, the patient is able and willing to comply with study visits and procedures (including laboratory tests, lung function tests).
* Subjects must be able to demonstrate ability to use salbutamol MDI during the screening period

Exclusion Criteria:

* The patient has currently poorly controlled disease defined as requiring a course of oral or parenteral corticosteroids or an exacerbation of their obstructive lung disease in the three months prior to Visit 2.
* The patient has had a recent change in maintenance therapy (i.e. within 6 weeks)
* Maintenance oral corticosteroid treatment or use of unlicensed doses of inhaled corticosteroid medication (>2000mcg beclomethasone diproprionate/ day or equivalent)
* The patient has seasonal disease alone
* The patient has any known laboratory abnormality, which in the opinion of the investigator, would contraindicate study participation, including, aspartate aminotransferase (AST) or alanine aminotransferase (ALT)greater/equal to 1.5 x upper limit of normal (ULN) or creatinine > 1.5 mg/dL
* The patient is unable to discontinue short-acting beta-2-adrenergic agonists for at least 4 hours, long-acting beta agonists (12 hours) and tiotropium (24 hours) prior to Visit 2 (Week 0)
* The patient has chronic heart failure class III or IV (New York Heart Association) or a recent (less than six months) history of stroke, transient ischemic attack or myocardial infarction
* The patient is not able to follow study procedures (e.g., language problems, psychological disorders) or is considered to be non-compliant according to the investigator.
* The patient has a history of known alcohol or substance abuse (excluding cigarettes) within the one-year prior to Visit 1
* The patient has an active malignancy of any type or history of a malignancy (with the exception of patients with malignancy surgically removed with no evidence of recurrence within five years before enrolment, and patients with history of treated basal cell carcinoma)
* The patient has any other severe or acute or chronic medical or psychiatric conditions that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study. Subjects with a malignancy and who are currently undergoing radiation therapy or have had chemotherapy within 5 years.
* The patient has difficulty swallowing capsules or tablets, dysphagia or is unable to tolerate oral medication
* The patient has been previously admitted to the study or currently participating or have recently participated in another trial with an investigational drug within 90 days of the start of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
The change in the Leicester Cough Questionnaire (LCQ) score | 8 weeks

SECONDARY OUTCOMES:
St Georges Respiratory Questionnaire (SGRQ) score | 8 weeks
EQ-5D score | 8 weeks
Spirometry (FEV1, FVC, PEF, FEF25-75 predicted) | 8 weeks
Impulse Oscillometry | 8 weeks
Differential spontaneous sputum cell count; TNFα,IL-8, IL-10 concentration | 8 weeks
Modified MRC dyspnoea score | 8 weeks
6 minute walk | 8 weeks
Blood haematology and biochemistry | 10 weeks
Drug related adverse events | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wilson, MD, MRCP (UK), Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Background] Tang Y, Xu Y, Xiong S, Ni W, Chen S, Gao B, Ye T, Cao Y, Du C. The effect of Ginkgo Biloba extract on the expression of PKCalpha in the inflammatory cells and the level of IL-5 in induced sputum of asthmatic patients. J Huazhong Univ Sci Technolog Med Sci. 2007 Aug;27(4):375-80. doi: 10.1007/s11596-007-0407-4. PMID 17828490
- [Background] Thomas M, Sheran J, Smith N, Fonseca S, Lee AJ. AKL1, a botanical mixture for the treatment of asthma: a randomised, double-blind, placebo-controlled, cross-over study. BMC Pulm Med. 2007 Mar 20;7:4. doi: 10.1186/1471-2466-7-4. PMID 17374147
- [Background] Birring SS, Prudon B, Carr AJ, Singh SJ, Morgan MD, Pavord ID. Development of a symptom specific health status measure for patients with chronic cough: Leicester Cough Questionnaire (LCQ). Thorax. 2003 Apr;58(4):339-43. doi: 10.1136/thorax.58.4.339. PMID 12668799
- [Background] Levy ML, Fletcher M, Price DB, Hausen T, Halbert RJ, Yawn BP. International Primary Care Respiratory Group (IPCRG) Guidelines: diagnosis of respiratory diseases in primary care. Prim Care Respir J. 2006 Feb;15(1):20-34. doi: 10.1016/j.pcrj.2005.10.004. Epub 2005 Dec 27. PMID 16701756
- [Background] Jones PW, Quirk FH, Baveystock CM, Littlejohns P. A self-complete measure of health status for chronic airflow limitation. The St. George's Respiratory Questionnaire. Am Rev Respir Dis. 1992 Jun;145(6):1321-7. doi: 10.1164/ajrccm/145.6.1321. PMID 1595997
- [Background] Dolan P. Modeling valuations for EuroQol health states. Med Care. 1997 Nov;35(11):1095-108. doi: 10.1097/00005650-199711000-00002. PMID 9366889
- [Background] van der Molen T, Willemse BW, Schokker S, ten Hacken NH, Postma DS, Juniper EF. Development, validity and responsiveness of the Clinical COPD Questionnaire. Health Qual Life Outcomes. 2003 Apr 28;1:13. doi: 10.1186/1477-7525-1-13. PMID 12773199
- [Background] Standardization of Spirometry, 1994 Update. American Thoracic Society. Am J Respir Crit Care Med. 1995 Sep;152(3):1107-36. doi: 10.1164/ajrccm.152.3.7663792. No abstract available.
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Background] Cote CG, Pinto-Plata V, Kasprzyk K, Dordelly LJ, Celli BR. The 6-min walk distance, peak oxygen uptake, and mortality in COPD. Chest. 2007 Dec;132(6):1778-85. doi: 10.1378/chest.07-2050. Epub 2007 Oct 9. PMID 17925409